CLINICAL TRIAL: NCT05125185
Title: The Effectiveness of USM-Insulin Adherence Module (U-IAM) for Type 2 Diabetes in Improving Insulin Adherence, Glycemic Control and Inflammation
Brief Title: The Effect of USM-IAM-based Counselling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Aida Maziha Binti Zainudin, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 304/PPSP/6315140
Record Dates: First submitted 2021-10-27; First posted 2021-11-18 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Type 2 on Insulin
MeSH Terms: interventions — Glycemic Control

STUDY DESIGN:
Intervention Model Description: comparing effect of counseling to insulin adherence, FBS, HbA1c, HsCRP and VCAM-1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Counseling (Active Comparator): Trained diabetic educators educate patients using flip charts produced based on Malaysian Diabetes educators' manuals, insulin pen models and handouts. All patients were given SMBG diaries and encouraged to titrate their insulin dose based on SMBG
  Interventions: Other: The Effectiveness of USM-Insulin Adherence Module (U-IAM) for Type 2 Diabetes in Improving Insulin Adherence, Glycemic Control and Inflammation
- USM-IAM- based counseling (Experimental): Trained diabetes educators counselled patients using the USM Insulin adherence module. Each patient was given the module so that they could freely refer to it when necessary. The module contains all information from standard counseling, with additional info on the definition of insulin non-adherence, causes of non-adherence, measures to overcome non-adherence and fasting safely with insulin. All patients were given SMBG diaries and encouraged to titrate their insulin dose based on SMBG
  Interventions: Other: The Effectiveness of USM-Insulin Adherence Module (U-IAM) for Type 2 Diabetes in Improving Insulin Adherence, Glycemic Control and Inflammation

INTERVENTIONS:
Other: The Effectiveness of USM-Insulin Adherence Module (U-IAM) for Type 2 Diabetes in Improving Insulin Adherence, Glycemic Control and Inflammation — To study the effect of counseling using USM-Insulin Adherence Module (U-IAM) for Type 2 Diabetes in improving Insulin Adherence, Glycemic Control and Inflammation

SUMMARY:
According to the most current local data, the rate of patient's adherence to insulin injections is very low. A recent cross sectional study in Klinik Pakar Perubatan (KPP) Hospital Universiti Sains Malaysia (HUSM) among 355 patients with Type 2 diabetes treated with insulin showed only 19% of patients adhered to their insulin regime with the mean fasting plasma glucose of 10mmol/L and mean HbA1C of 10.0%. This condition may lead to undesirable health consequences.

Patients education has been showed to improved adherence. Among the 355 participants involved in the study, 82% of the patients have received consultation by diabetic educators yet their glycemic control were suboptimal. A new approaches using a module-based counseling that emphasized on adherence has been developed and the effectiveness of the counseling need to be evaluated.

DETAILED DESCRIPTION:
General objective: To determine the effect of USM-insulin adherence module (U-IAM)-based counseling on the insulin adherence, glycemic control and inflammatory markers in poorly-controlled type 2 diabetes mellitus patients on insulin therapy.

Specific objective:

1. To determine within group changes and between group differences of insulin adherence score (using IAQDM) between patients in intervention and control group at baseline, 3rd month and 6th month
2. To determine within group changes and between group differences of FBS and HbA1c between patients in intervention and control group at baseline, 3rd month and 6th month.
3. To determine within group changes and between group differences of HsCRP and VCAM-1 between patients in intervention and control group at baseline, 3rd month and 6th month.
4. To identify factors associated with nonadherence (before starting of intervention) among patients on insulin such as sociodemographic, SMBG and treatment factors.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 65 years
* have been diagnosed with Type 2 Diabetes Mellitus
* Patients treated with insulin injections for at least 1 year on either basal insulin, basal plus prandial or basal bolus insulin
* HbA1c between 8 % and 15%

Exclusion Criteria:

* do not understand Malay language or illiterate
* have severe diabetes complications such as chronic kidney disease, heart failure
* recurrent hypoglycemia or hypoglycemia unawareness
* body mass index (BMI) ≥ 40kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change of insulin adherence score | 3 months
  Insulin adherence will be measured using an insulin adherence questionnaire for diabetes. change from mellitus. It contains 34 questions with minimum marks of 0 and a maximum of 100 marks. The higher the marks, the higher the degree of adherence. The patient is considered to adhere if they achieved marks of equal or more than 80
Change of insulin adherence score | 6 months
  Insulin adherence will be measured using insulin adherence questionnaire for diabetes mellitus. it contains 34 questions with minimum marks of 0 and maximum of 100 marks. The higher the marks, the higher the degree of adherence. Patient is considered adherence if they achieved marks of equal or more than 80
Change of Fasting Blood Sugar | 3 months
  change of FBS from baseline to 3 months
Change of Fasting Blood Sugar | 6 months
  change of FBS from baseline to 6 months
Change of HbA1c | 3 months
  change of HbA1c from baseline to 3 months
Change of HbA1c | 6 months
  change of HbA1c from baseline to 6 months
Change of HsCRP | 6 months
  change of HsCRP from baseline to 6 months
Change of VCAM-1 | 6 months
  change of baseline from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aida Maziha Zainudin, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

REFERENCES:
- [Derived] Zainudin AM, Rasool AHG, Yaacob NM, Muhamad R, Mohamed WMIW. The effect of USM-IAM-based counselling vs standard counselling on insulin adherence, FBS and HbA1c among patients with uncontrolled type 2 diabetes mellitus (T2DM): a randomised controlled trial. BMC Endocr Disord. 2024 Jul 18;24(1):118. doi: 10.1186/s12902-024-01577-6. PMID 39020348